CLINICAL TRIAL: NCT03253939
Title: Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy in Peritoneal Carcinomatosis From Gastric Cancer
Acronym: CYTO-CHIP
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CYTO-CHIP
Record Dates: First submitted 2017-07-27; First posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-07

CONDITIONS: Gastric Cancer; Peritoneal Carcinomatosis
MeSH Terms: conditions — Stomach Neoplasms; Peritoneal Neoplasms | interventions — Cytoreduction Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy procedure
  Interventions: Procedure: Cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy procedure
- Control group: Cytoreductive surgery alone
  Interventions: Procedure: Cytoreductive surgery alone

INTERVENTIONS:
Procedure: Cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy procedure — Cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy procedure
  Groups: Case group
Procedure: Cytoreductive surgery alone — Exclusively Cytoreductive surgery approach
  Groups: Control group

SUMMARY:
Gastric cancer associated peritoneal carcinomatosis has a poor prognosis with a median survival of less than one year. Systemic chemotherapy including targeted agents has not been found to significantly increase the survival in Gastric cancer associated peritoneal carcinomatosis. Since recurrent gastric cancer remains confined to the abdominal cavity in many patients, regional therapies like aggressive cytoreductive surgery and hyperthermic intraperitoneal chemotherapy have been investigated for Gastric cancer associated peritoneal carcinomatosis. Hyperthermic intraperitoneal chemotherapy has been used for three indications in Gastric Cancer- as an adjuvant therapy after a curative surgery, hyperthermic intraperitoneal chemotherapy has been shown to improve survival and reduce peritoneal recurrences in many randomised trials in Asian countries; as a definitive treatment in established PC, hyperthermic intraperitoneal chemotherapy along with cytoreductive surgery is the only therapeutic modality that has resulted in long-term survival in select groups of patients. While the results of randomised trials of adjuvant hyperthermic intraperitoneal chemotherapy from western centres are awaited, the role of hyperthermic intraperitoneal chemotherapy in the treatment of Gastric cancer associated peritoneal carcinomatosis is still evolving and needs larger studies before it is accepted as a standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed peritoneal carcinomatosis from gastric cancer
* Metachronous/synchronous peritoneal carcinomatosis

Exclusion Criteria:

- Gastric origin of peritoneal carcinomatosis unconfirmed

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastric peritoneal carcinomatosis. All patients received the current standard neoadjuvant treatment.
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
3-years overall survival | 3 years
  From the date of Cytoreductive surgery + hyperthermic intraperitoneal chemotherapy to death or to the end of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Générale et Digestive - Centre Hospitalier Lyon Sud - Hospices Civils de Lyon, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bonnot PE, Piessen G, Kepenekian V, Decullier E, Pocard M, Meunier B, Bereder JM, Abboud K, Marchal F, Quenet F, Goere D, Msika S, Arvieux C, Pirro N, Wernert R, Rat P, Gagniere J, Lefevre JH, Courvoisier T, Kianmanesh R, Vaudoyer D, Rivoire M, Meeus P, Passot G, Glehen O; FREGAT and BIG-RENAPE Networks. Cytoreductive Surgery With or Without Hyperthermic Intraperitoneal Chemotherapy for Gastric Cancer With Peritoneal Metastases (CYTO-CHIP study): A Propensity Score Analysis. J Clin Oncol. 2019 Aug 10;37(23):2028-2040. doi: 10.1200/JCO.18.01688. Epub 2019 May 14. PMID 31084544